CLINICAL TRIAL: NCT03491072
Title: Transcutaneous Electric Nerve Stimulation (TENS) for Pain Relief During Extracorporeal Shock-wave Lithotripsy (ESWL)
Brief Title: Transcutaneous Electric Nerve Stimulation for Pain Relief During Extracorporeal Shock-wave Lithotripsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Randa Ali Shoukry, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R 12/2018
Record Dates: First submitted 2018-03-31; First posted 2018-04-09 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Pain
Keywords: extracorporeal shock-wave Lithotripsy,; pain relief during extracorporeal shock-wave Lithotripsy; fentanyl; Transcutaneous electrical nerve stimulation
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation; Fentanyl; Injections, Intravenous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous electrical nerve stimulation (TENS) (Experimental): Patients will receive IV fentanyl 1µg /Kg with the application of conventional TENS in which constant mode will be chosen. Assessment of pain will be done using visual analogue scale (VAS), every 10 minutes. If VAS ≥ 3 this indicates giving IV increments of 20µg of fentanyl.
  Interventions: Device: Transcutaneous electrical nerve stimulation; Drug: Fentanyl
- Fentanyl (Active Comparator): Patients will receive IV fentanyl 1µg /Kg. Assessment of pain will be done using visual analogue scale (VAS), every 10 minutes. If VAS ≥ 3 this indicates giving IV increments of 20µg of fentanyl.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation — Patients will receive IV fentanyl 1µg /Kg with the application of conventional TENS in which constant mode will be chosen. Assessment of pain will be done using visual analogue scale (VAS), every 10 minutes. If VAS ≥ 3 this indicates giving IV increments of 20µg of fentanyl.
  Other Names: TENS
  Arms: Transcutaneous electrical nerve stimulation (TENS)
Drug: Fentanyl — Patients will receive IV fentanyl
  Other Names: Fentanyl ampule for intravenous injection

SUMMARY:
This study evaluates pain relief during extracorporeal shock-wave Lithotripsy by using transcutaneous electrical nerve stimulation (TENS) and comparing it with fentanyl which is a narcotic analgesic. Half of the participants will receive a primary fentanyl dose together with TENS application, another half will receive a primary fentanyl dose. All patients will receive fentanyl increments if they still complained of pain.

DETAILED DESCRIPTION:
The ideal anesthesia technique for ESWL must provide good analgesia, sufficient sedation, and rapid recovery with minimal side effects. Opioids are commonly used analgesics during ESWL. Fentanyl is a potent synthetic narcotic, which has rapid onset and a short duration of action, it offers an acceptable analgesia during ESWL but has a noticeable respiratory depression.

Transcutaneous electrical nerve stimulation (TENS) is a method in which low voltage electrical impulses transmit through electrodes attached to the skin over a painful area. It is usually used to relieve a variety of painful conditions. A TENS unit contains electrical signal generator, a battery in addition to a set of electrodes. The TENS is small, programmable and the generator can deliver stimuli with different current intensities, pulse rates and pulse width.

The mechanism of analgesia by TENS has been explained by many theories. the gate control theory by Melzack and Wall, stated that "when an electrical current is applied to a painful area, transmission of pain through small diameter fibers is inhibited by the activity of the large diameter, fast-conducting proprioceptive sensory fibers, closing the gate to the pain perception to the brain". Another mechanism suggested is activation of descending inhibitory pathway, via release of endogenous opioids.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for extracorporeal shock-wave Lithotripsy (ESWL), having a solitary renal stone 6 - 15 mm.
* Age18 to 75 years old.
* ASA physical status I -II.
* BMI of 25- 30.

Exclusion Criteria:

* Patients with bleeding and coagulation disorder.
* Hypertension.
* Pregnancy,
* Patient with demand pacemaker.
* Dermatological lesions at the site of ESWL e.g. eczema or dermatitis.
* Drug or alcohol addiction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Pain intensity measure using visual analogue scale | 10 minutes
  patients will be instructed to mark the line with a pencil (0 = no pain 10= worst pain).

SECONDARY OUTCOMES:
Fentanyl consumption | during the procedure of ESWL
  Total dose of requested and received fentanyl.

CONTACTS AND LOCATIONS:
Overall Officials: Randa AS Ahmed, MD, Principal Investigator — Ain Shams University
Locations (1):
- Randa Ali Shoukry, Cairo, Al-Nozha, Egypt